CLINICAL TRIAL: NCT07002736
Title: The Impact of Balance Training on Functional Performance and Fall Risk in Community-Dwelling Older Adults Following Recovery From COVID-19"
Brief Title: Impact of Balance Training in Community-Dwelling Older Adults After Recovery From COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mariam Elsayed Mohamed Abd Alaal, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Balance and covid 19
Record Dates: First submitted 2025-06-01; First posted 2025-06-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-06

CONDITIONS: Community-dwelling Older Adults
Keywords: older adults; Berg Balance Scale; COVID-19; Biodex
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Biodex training (Experimental): Balance Training
  Interventions: Other: The Biodex training; Other: Traditional balance training
- Control (Active Comparator): Traditional Balance Training
  Interventions: Other: Traditional balance training

INTERVENTIONS:
Other: The Biodex training — Participants will undergo balance training using the Biodex Balance System plus Traditional balance training
  Arms: The Biodex training
Other: Traditional balance training — Traditional balance training only

SUMMARY:
This research investigates the impact of balance training on improving functional performance and reducing fall risk in community-dwelling older adults who have recovered from COVID-19. Post-COVID-19, many elderly individuals experience lingering physical impairments, including muscle weakness, decreased coordination, and balance deficits, which increase their vulnerability to falls. The study evaluates whether a structured balance training program can enhance stability, mobility, and overall quality of life in this population.

DETAILED DESCRIPTION:
Older adults recovering from COVID-19 frequently face persistent physical limitations due to the virus's impact on the respiratory, muscular, and neurological systems. These limitations often manifest as impaired balance, reduced functional mobility, and increased risk of falls-conditions further exacerbated by prolonged inactivity or hospitalization during illness.

This research focuses on evaluating the effectiveness of a structured balance training program using The Biodex Stability System in older adults living independently in the community after recovering from COVID-19.

Participants are assessed using validated tools such as the Berg Balance Scale, Timed Up and Go (TUG) test, and The Biodex Stability System to measure changes in balance performance, fall risk, and confidence in daily movement.

ELIGIBILITY:
Inclusion Criteria:

* were being older adults (aged ≥60 years), recovered from infection during the last 6 month,

Exclusion Criteria:

* Individuals were excluded if they have medical history of musculoskeletal trauma or surgery, systemic disease that could affect standing or walking, visual, auditory, or cognitive impairment that preclude the ability to comprehend the instructions during conduction of the study protocol.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Biodex Balance indices | Pre and Post 12 weeks
  The Biodex Stability System will be used to evaluate dynamic postural stability
Berg Balance Scale score | Pre and Post 12 weeks
  The Berg Balance Scale will be used to evaluate balance capability

SECONDARY OUTCOMES:
Timed up and Go test | Pre and Post 12 weeks
  Timed up and Go test will be used to assess functional mobility, dynamic balance, and fall risk in older adults

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mariam Salem, Principal Investigator — BMC
Locations (1):
- BMC, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Bagalaty AE, Mohamed ME, Abdelraouf OR, Abdel Ghafar MA, Abdelaal AK, Abdelgalil AA, Mousa GS. Balance and Fall Risk Assessment in Community-Dwelling Older Adults after Recovery from COVID-19: A Cross-Sectional Study. Sports (Basel). 2023 Jan 28;11(2):28. doi: 10.3390/sports11020028. PMID 36828313